CLINICAL TRIAL: NCT03198871
Title: Role of Scheduled Intravenous Acetaminophen for Postoperative Pain Management in an Enhanced Recovery After Surgery (ERAS) Population: A Prospective, Randomized, Double-Blind and Placebo-Controlled Clinical Trial
Brief Title: IV Acetaminophen for Post-Operative Pain Management in Enhanced Recovery After Surgery (ERAS) Population
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kathirvel Subramaniam (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Sponsor-Investigator, Kathirvel Subramaniam, Principal Investigator, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRO17050418
Record Dates: First submitted 2017-06-19; First posted 2017-06-26 (Actual); Results first posted 2021-01-28 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Abdominal Wall Hernia; Pancreatic Diseases; Bowel Disease; Gastric Disease
Keywords: Post-operative pain; Major abdominal surgery; Colorectal surgery; Gastric surgery
MeSH Terms: conditions — Hernia, Abdominal; Pancreatic Diseases; Intestinal Diseases; Stomach Diseases; Pain, Postoperative | interventions — Acetaminophen; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participant, care provider, outcomes assessor and investigator are all blinded to the treatment allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Acetaminophen Injectable Product (Experimental): Acetaminophen group: Half of subjects enrolled will be randomized to the acetaminophen group
  Interventions: Drug: Acetaminophen Injectable Product
- Sodium Chloride 0.9%, Intravenous (Placebo Comparator): Sodium Chloride 0.9% group: Half of subjects enrolled will be randomized to the acetaminophen group
  Interventions: Drug: Sodium Chloride 0.9%, Intravenous

INTERVENTIONS:
Drug: Acetaminophen Injectable Product — The interventional group will receive 1 gram intravenous acetaminophen at the start of wound closure to be repeated every 6 hours for 48 hours postoperatively
  Other Names: Tylenol; Paracetamol; Ofirmev
  Arms: Acetaminophen Injectable Product
Drug: Sodium Chloride 0.9%, Intravenous — The placebo group will be given an intravenous placebo of saline solution at wound closure and repeated every 6 hours for 48 hours postoperatively.
  Other Names: Saline
  Arms: Sodium Chloride 0.9%, Intravenous

SUMMARY:
Number of patients with unsatisfactory pain relief defined as average visual analog scale (VAS) more than 5 with or without requirement of IVPCA for pain relief during the first 48 hours postoperative period will be compared between the two groups and form the primary outcome for the study. Postoperative pain intensity will be measured by Visual Analog Scale (VAS) with 0- being no pain and 10-being maximum pain and the analgesic efficacy in both groups will also be evaluated by the amount of total narcotic consumption (measured with IV morphine equivalent doses of analgesics used to provide pain relief).

DETAILED DESCRIPTION:
In response to an increased focus on improving patient outcomes and satisfaction with surgical care, a growing body of clinical evidence has recently been dedicated to enhanced recovery after surgery (ERAS) protocols. These evidence-based perioperative pathways aim to optimize patients undergoing surgery in the preoperative, intraoperative, and postoperative periods. ERAS protocols have incorporated the use of multimodal analgesia to minimize the use of intra- and postoperative opioid analgesics. Lidocaine, ketamine, magnesium, gabapentin, acetaminophen and non-steroidal anti-inflammatory drugs are some of the adjuvant analgesics used in combination with regional blocks to optimize analgesia and recovery. Multimodal analgesia has dependably been shown to significantly reduce postoperative opioid requirements as well as opioid-related side effects such as postoperative nausea and vomiting. Both oral and intravenous acetaminophen preparations have been shown to be useful adjuvants in multimodal analgesia. Intravenous acetaminophen has been of interest for its utility in post-surgical patients, who have not yet been cleared for oral intake. Intravenous acetaminophen should also be preferred over oral acetaminophen in patients after major abdominal surgery where absorption of medications given through oral route is erratic. Although the efficacy of intravenous acetaminophen as a postoperative pain adjunct is known, its exact role in ERAS protocols and non-narcotic multimodal analgesic regimens for major abdominal surgery has not been studied in randomized clinical trials to define its efficacy. The primary goal of this study is to assess the utility of a postoperative intravenous acetaminophen dosing schedule in minimizing postoperative pain, opioid consumption and opioid-related side effects. We also aim to study overall patient satisfaction and cost-effectiveness (direct and indirect costs) of this regimen as part of ERAS protocol at a large tertiary medical center.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* 18 years of age or older
* patients scheduled for elective colorectal, pancreatic, and other major abdominal procedure.
* Patient consent will be obtained preoperatively for eligible study participants.

Exclusion Criteria:

* Patients who refuse to participate in the study or part of any other enhanced recovery after surgery (ERAS) research protocol.
* Patients with a documented allergy to acetaminophen.
* Chronic alcoholism
* Hypovolemia
* Chronic malnutrition
* Preoperative renal insufficiency (creatinine clearance less than or equal to 30ml/min) or hemodialysis
* Patients with a history of hepatic impairment, history of hepatic impairment or active hepatic disease
* severe chronic pain condition that required daily preoperative opioid dependence
* Patients with pre-existing dementia and/or other neuropsychiatric conditions impeding accurate assessment of pain scores or other study measures will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2018-05-24 (Actual); Primary Completion 2019-07-07 (Actual); Study Completion 2020-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathirvel Subramaniam, M.D., M.P.H, Principal Investigator — Associate Professor and staff Anesthesiologist
Locations (1):
- Upmc Presbyterian Montefiore Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ziemann-Gimmel P, Hensel P, Koppman J, Marema R. Multimodal analgesia reduces narcotic requirements and antiemetic rescue medication in laparoscopic Roux-en-Y gastric bypass surgery. Surg Obes Relat Dis. 2013 Nov-Dec;9(6):975-80. doi: 10.1016/j.soard.2013.02.003. Epub 2013 Feb 13. PMID 23499469
- [Background] Ziemann-Gimmel P, Goldfarb AA, Koppman J, Marema RT. Opioid-free total intravenous anaesthesia reduces postoperative nausea and vomiting in bariatric surgery beyond triple prophylaxis. Br J Anaesth. 2014 May;112(5):906-11. doi: 10.1093/bja/aet551. Epub 2014 Feb 18. PMID 24554545
- [Background] Practice guidelines for acute pain management in the perioperative setting. A report by the American Society of Anesthesiologists Task Force on Pain Management, Acute Pain Section. Anesthesiology. 1995 Apr;82(4):1071-81. No abstract available. PMID 7717542
- [Background] Hansen RN, Pham A, Strassels SA, Balaban S, Wan GJ. Erratum to: Comparative Analysis of Length of Stay and Inpatient Costs for Orthopedic Surgery Patients Treated with IV Acetaminophen and IV Opioids vs. IV Opioids Alone for Post-Operative Pain. Adv Ther. 2016 Sep;33(9):1646-1648. doi: 10.1007/s12325-016-0400-z. No abstract available. PMID 27562836
- [Background] Bollinger AJ, Butler PD, Nies MS, Sietsema DL, Jones CB, Endres TJ. Is Scheduled Intravenous Acetaminophen Effective in the Pain Management Protocol of Geriatric Hip Fractures? Geriatr Orthop Surg Rehabil. 2015 Sep;6(3):202-8. doi: 10.1177/2151458515588560. PMID 26328237
- [Background] Herring BO, Ader S, Maldonado A, Hawkins C, Kearson M, Camejo M. Impact of intravenous acetaminophen on reducing opioid use after hysterectomy. Pharmacotherapy. 2014 Dec;34 Suppl 1:27S-33S. doi: 10.1002/phar.1513. PMID 25521844
- [Background] Jokela R, Ahonen J, Seitsonen E, Marjakangas P, Korttila K. The influence of ondansetron on the analgesic effect of acetaminophen after laparoscopic hysterectomy. Clin Pharmacol Ther. 2010 Jun;87(6):672-8. doi: 10.1038/clpt.2009.281. Epub 2010 Mar 10. PMID 20220746
- [Background] Gonzalez A, Ziemann-Gimmel P. The role of multimodal analgesia in bariatric surgery: A review of clinical data and case-based presentations featuring OFIRMEV® (acetaminophen) injection. Surgical Pain Management. 2014;11(5): A2-11.
- [Background] Pettersson PH, Jakobsson J, Owall A. Intravenous acetaminophen reduced the use of opioids compared with oral administration after coronary artery bypass grafting. J Cardiothorac Vasc Anesth. 2005 Jun;19(3):306-9. doi: 10.1053/j.jvca.2005.03.006. PMID 16130055
- [Background] Mamoun NF, Lin P, Zimmerman NM, Mascha EJ, Mick SL, Insler SR, Sessler DI, Duncan AE. Intravenous acetaminophen analgesia after cardiac surgery: A randomized, blinded, controlled superiority trial. J Thorac Cardiovasc Surg. 2016 Sep;152(3):881-889.e1. doi: 10.1016/j.jtcvs.2016.04.078. Epub 2016 May 5. PMID 27236864
- [Background] Douzjian DJ, Kulik A. Old Drug, New Route: A Systematic Review of Intravenous Acetaminophen After Adult Cardiac Surgery. J Cardiothorac Vasc Anesth. 2017 Apr;31(2):694-701. doi: 10.1053/j.jvca.2016.03.134. Epub 2016 Mar 16. No abstract available. PMID 27498260
- [Background] Thiele RH, Rea KM, Turrentine FE, Friel CM, Hassinger TE, McMurry TL, Goudreau BJ, Umapathi BA, Kron IL, Sawyer RG, Hedrick TL. Standardization of care: impact of an enhanced recovery protocol on length of stay, complications, and direct costs after colorectal surgery. J Am Coll Surg. 2015 Apr;220(4):430-43. doi: 10.1016/j.jamcollsurg.2014.12.042. Epub 2015 Jan 9. PMID 25797725
- [Background] Doleman B, Read D, Lund JN, Williams JP. Preventive Acetaminophen Reduces Postoperative Opioid Consumption, Vomiting, and Pain Scores After Surgery: Systematic Review and Meta-Analysis. Reg Anesth Pain Med. 2015 Nov-Dec;40(6):706-12. doi: 10.1097/AAP.0000000000000311. PMID 26469366
- [Background] Remy C, Marret E, Bonnet F. Effects of acetaminophen on morphine side-effects and consumption after major surgery: meta-analysis of randomized controlled trials. Br J Anaesth. 2005 Apr;94(4):505-13. doi: 10.1093/bja/aei085. Epub 2005 Jan 28. PMID 15681586
- [Background] Macario A, Royal MA. A literature review of randomized clinical trials of intravenous acetaminophen (paracetamol) for acute postoperative pain. Pain Pract. 2011 May-Jun;11(3):290-6. doi: 10.1111/j.1533-2500.2010.00426.x. Epub 2010 Nov 28. PMID 21114616
- [Background] Cakan T, Inan N, Culhaoglu S, Bakkal K, Basar H. Intravenous paracetamol improves the quality of postoperative analgesia but does not decrease narcotic requirements. J Neurosurg Anesthesiol. 2008 Jul;20(3):169-73. doi: 10.1097/ANA.0b013e3181705cfb. PMID 18580346
- [Background] Brett CN, Barnett SG, Pearson J. Postoperative plasma paracetamol levels following oral or intravenous paracetamol administration: a double-blind randomised controlled trial. Anaesth Intensive Care. 2012 Jan;40(1):166-71. doi: 10.1177/0310057X1204000121. PMID 22313079
- [Background] Fenlon S, Collyer J, Giles J, Bidd H, Lees M, Nicholson J, Dulai R, Hankins M, Edelman N. Oral vs intravenous paracetamol for lower third molar extractions under general anaesthesia: is oral administration inferior? Br J Anaesth. 2013 Mar;110(3):432-7. doi: 10.1093/bja/aes387. Epub 2012 Dec 6. PMID 23220855
- [Background] Wang S, Saha R, Shah N, Hanna A, DeMuro J, Calixte R, Brathwaite C. Effect of Intravenous Acetaminophen on Postoperative Opioid Use in Bariatric Surgery Patients. P T. 2015 Dec;40(12):847-50. PMID 26681907
- [Background] Bameshki A, Peivandi Yazdi A, Sheybani S, Rezaei Boroujerdi H, Taghavi Gilani M. The Assessment of Addition of Either Intravenous Paracetamol or Diclofenac Suppositories to Patient-Controlled Morphine Analgesia for Postgastrectomy Pain Control. Anesth Pain Med. 2015 Oct 10;5(5):e29688. doi: 10.5812/aapm.29688. eCollection 2015 Oct. PMID 26587407
- [Background] Strode MA, Sherman W, Mangieri CW, Bland CM, Sparks PJ, Faler BJ, Prasad BM, Choi YU. Randomized trial of OFIRMEV versus placebo for pain management after laparoscopic sleeve gastrectomy. Surg Obes Relat Dis. 2016 May;12(4):772-777. doi: 10.1016/j.soard.2015.08.512. Epub 2015 Aug 29. PMID 26525369
- [Background] Saurabh S, Smith JK, Pedersen M, Jose P, Nau P, Samuel I. Scheduled intravenous acetaminophen reduces postoperative narcotic analgesic demand and requirement after laparoscopic Roux-en-Y gastric bypass. Surg Obes Relat Dis. 2015 Mar-Apr;11(2):424-30. doi: 10.1016/j.soard.2014.09.017. Epub 2014 Sep 30. PMID 25614351
- [Background] Song K, Melroy MJ, Whipple OC. Optimizing multimodal analgesia with intravenous acetaminophen and opioids in postoperative bariatric patients. Pharmacotherapy. 2014 Dec;34 Suppl 1:14S-21S. doi: 10.1002/phar.1517. PMID 25521841
- [Background] Ziolkowski K, Kaufman J, Jambunathan J, Berge J, Menet L, Chappy S, Messerschmidt M. The Clinical Use of Intravenous Acetaminophen Postoperatively on Patients Who Have Undergone Bowel Surgery. AORN J. 2015 Nov;102(5):515.e1-515.e10. doi: 10.1016/j.aorn.2015.09.011. PMID 26514714
- [Background] Wininger SJ, Miller H, Minkowitz HS, Royal MA, Ang RY, Breitmeyer JB, Singla NK. A randomized, double-blind, placebo-controlled, multicenter, repeat-dose study of two intravenous acetaminophen dosing regimens for the treatment of pain after abdominal laparoscopic surgery. Clin Ther. 2010 Dec;32(14):2348-69. doi: 10.1016/j.clinthera.2010.12.011. PMID 21353105
- [Background] Apfel CC, Turan A, Souza K, Pergolizzi J, Hornuss C. Intravenous acetaminophen reduces postoperative nausea and vomiting: a systematic review and meta-analysis. Pain. 2013 May;154(5):677-689. doi: 10.1016/j.pain.2012.12.025. Epub 2013 Jan 11. PMID 23433945
- [Background] Guha A, Scawn ND, Rogers SA, Pennefather SH, Russell GN. Gastric emptying in post-thoracotomy patients receiving a thoracic fentanyl-bupivacaine epidural infusion. Eur J Anaesthesiol. 2002 Sep;19(9):652-7. doi: 10.1017/s0265021502001072. PMID 12243288
- [Background] Yuan CS, Foss JF, O'Connor M, Roizen MF, Moss J. Effects of low-dose morphine on gastric emptying in healthy volunteers. J Clin Pharmacol. 1998 Nov;38(11):1017-20. doi: 10.1177/009127009803801105. PMID 9824782
- [Background] Jibril F, Sharaby S, Mohamed A, Wilby KJ. Intravenous versus Oral Acetaminophen for Pain: Systematic Review of Current Evidence to Support Clinical Decision-Making. Can J Hosp Pharm. 2015 May-Jun;68(3):238-47. doi: 10.4212/cjhp.v68i3.1458. PMID 26157186
- [Background] El Chaar M, Stoltzfus J, Claros L, Wasylik T. IV Acetaminophen Results in Lower Hospital Costs and Emergency Room Visits Following Bariatric Surgery: a Double-Blind, Prospective, Randomized Trial in a Single Accredited Bariatric Center. J Gastrointest Surg. 2016 Apr;20(4):715-24. doi: 10.1007/s11605-016-3088-0. Epub 2016 Feb 2. PMID 26842692
- [Background] Apfel CC, Souza K, Portillo J, Dalal P, Bergese SD. Patient satisfaction with intravenous acetaminophen: a pooled analysis of five randomized, placebo-controlled studies in the acute postoperative setting. J Healthc Qual. 2015 May-Jun;37(3):155-62. doi: 10.1111/jhq.12062. PMID 24433365
- [Derived] Subramaniam K, Esper SA, Mallikarjun K, Dickson A, Ruppert DrPH K, Drabek T, Wong H, Holder-Murray J. The Effect of Scheduled Intravenous Acetaminophen in an Enhanced Recovery Protocol Pathway in Patients Undergoing Major Abdominal Procedures: A Prospective, Randomized, and Placebo-Controlled Clinical Trial. Pain Med. 2022 Jan 3;23(1):10-18. doi: 10.1093/pm/pnab272. PMID 34498068

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Acetaminophen Injectable Product | Sodium Chloride 0.9%, Intravenous
Started | 90 | 90
Completed | 76 | 78
Not Completed | 14 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acetaminophen Injectable Product | Sodium Chloride 0.9%, Intravenous | Total
Number analyzed (Participants) | 76 | 78 | 154
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 62 [55 to 70.75] | 64 [53.75 to 74] | 63 [52.25 to 72.75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 44 | 84
  Male | 36 | 34 | 70
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 70 | 73 | 143
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 76 | 78 | 154
Basal Metabolic Index [Median (Inter-Quartile Range); unit: kg/m^2] | 27.7 [24.4 to 32.55] | 28.25 [23.8 to 32.4] | 28.15 [23.86 to 32.4]
Charlson Comorbidity Index [Count of Participants; unit: Participants] — 1 = Myocardial infarction history, CHF, PVD (aortic aneurism ≥6 cm), cerebrovascular disease: cerebrovascular accident +/- transient ischaemic attack, dementia, CPD, connective tissue disease, peptic ulcer disease, mild liver disease (w/o portal hypertension, includes chronic hepatitis), diabetes w/o end-organ damage (excludes diet-controlled) 2 = Hemiplegia, moderate/severe renal disease, diabetes w/ end-organ damage, tumour w/o metastases (<5 years from diagnosis), leukaemia, lymphoma 3 = Moderate/severe liver disease 6 = Metastatic solid tumour, AIDS. Add 1 for each decade >40yr.
  Participants
    0 | 44 | 41 | 85
    1 | 4 | 10 | 14
    2 | 23 | 24 | 47
    >2 | 5 | 3 | 8
American Society of Anesthesiologists Classification [Count of Participants; unit: Participants] — I = Healthy patients II = Mild to moderate systemic disease caused by the surgical condition or by other pathological processes, and medically well controlled III = Severe disease process which limits activity but is not incapacitating IV = Severe incapacitating disease process that is a constant threat to life V = Moribund patient not expected to survive 24 hours with or without an operation VI = Declared brain-dead patient whose organs are being removed for donor purposes
  Participants
    II | 17 | 18 | 35
    III | 57 | 55 | 112
    IV | 2 | 5 | 7
Number of participants taking medications for mental health [Count of Participants; unit: Participants] | 15 | 27 | 42
Diabetes [Count of Participants; unit: Participants] | 4 | 3 | 7
Hypertension [Count of Participants; unit: Participants] | 10 | 16 | 26
Coronary artery disease [Count of Participants; unit: Participants] | 2 | 4 | 6
Congestive failure [Count of Participants; unit: Participants] | 1 | 3 | 4
Atrial fibrillation [Count of Participants; unit: Participants] | 2 | 2 | 4
Pulmonary disease [Count of Participants; unit: Participants] | 3 | 6 | 9
Malignancy [Count of Participants; unit: Participants] | 28 | 23 | 51
Preoperative serum creatinine [Median (Inter-Quartile Range); unit: (mg/dL)] | 0.8 [0.7 to 1.0] | 0.82 [0.7 to 1.05] | 0.81 [0.7 to 1.0]

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Pain Intensity
Description: Number of patients with unsatisfactory pain relief defined as average numeric rating scale (NRS) more than 5 will be compared between the two groups. This may include patients using IVPCA for pain relief during the first 48 hours postoperative.
Time Frame: PACU admission every thirty minutes until discharge to the floor and thereafter every four hours for first 24-hour, then every six hours until 48 hours and then every twelve hours until 72 hours postoperatively.
Measure: Count of Participants; unit: Participants
Arm/Group | Acetaminophen Injectable Product | Sodium Chloride 0.9%, Intravenous
Number analyzed (Participants) | 76 | 78
Participants | 33 | 42

2. Secondary Outcome: Total Post-operative Narcotic Consumption
Description: Rescue analgesia will be given according to institutional pain management protocol. Unit of Measure recorded as OME (Oral Morphine Equivalent) consumption in mg.
Time Frame: From time of PACU admission until the time of discharge and 72-hours postoperatively, whichever comes first
Measure: Median (Inter-Quartile Range); unit: mg
Arm/Group | Acetaminophen Injectable Product | Sodium Chloride 0.9%, Intravenous
Number analyzed (Participants) | 76 | 78
mg
  0-24 hours | 27.4 [10 to 49] | 36 [17.5 to 85]
  24-48 hours | 31.3 [7.5 to 73.3] | 45 [15 to 95]
  48-72 hours | 30 [0 to 70] | 37.5 [0 to 70]
  0-48 hours | 74 [25.5 to 113] | 88.8 [42.5 to 167.5]
  0-72 hours | 105.00 [41.3 to 186.3] | 127.1 [49.3 to 252.00]

3. Secondary Outcome: Time to Readiness for Discharge From Post Anesthesia Care Unit (PACU)
Description: The time from PACU admission to PACU discharge to the floor will be measured.
Time Frame: From time of PACU admission until the time of discharge, assessed up to 24 hours postoperatively
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Acetaminophen Injectable Product | Sodium Chloride 0.9%, Intravenous
Number analyzed (Participants) | 76 | 78
minutes | 129.00 [106 to 186] | 152.50 [98.50 to 208.50]

4. Secondary Outcome: Time to Bowel Movement
Description: The time it takes for the first bowel movement postoperatively will be measured.
Time Frame: From time patient left operating room until the time of first documented bowel movement, assessed up to hospital discharge
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Acetaminophen Injectable Product | Sodium Chloride 0.9%, Intravenous
Number analyzed (Participants) | 76 | 78
hours | 46.30 [25.38 to 90.85] | 64.66 [29.27 to 115.33]

5. Secondary Outcome: Time to Oral Intake
Description: The time it takes for the patient to ingest orally post-surgery will be measured.
Time Frame: From date of randomization until the date of first documented oral intake, assessed up to 72 hours postoperatively
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Acetaminophen Injectable Product | Sodium Chloride 0.9%, Intravenous
Number analyzed (Participants) | 76 | 78
hours | 12.15 [4.53 to 33.17] | 9.40 [3.87 to 43.38]

6. Secondary Outcome: Time to Ambulation
Description: The time it takes for the patient to successfully ambulate post-surgery will be measured.
Time Frame: From date of PACU admission until the date of first documented ambulation, assessed up to 72 hours postoperatively
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Acetaminophen Injectable Product | Sodium Chloride 0.9%, Intravenous
Number analyzed (Participants) | 76 | 78
hours | 18.82 [4.42 to 37.77] | 17.38 [4.28 to 22.65]

7. Secondary Outcome: Time to Hospital Discharge
Description: The time it takes for the patient to be fully discharged from the hospital post-surgery will be measured.
Time Frame: From date of randomization until the date of hospital discharge or 30 days postoperatively, whichever comes first
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Acetaminophen Injectable Product | Sodium Chloride 0.9%, Intravenous
Number analyzed (Participants) | 76 | 78
days | 4.08 [3.07 to 6.04] | 4.94 [3.94 to 7.12]

8. Secondary Outcome: Number of Participants With Readmission to the Hospital
Description: If the patient is readmitted to the hospital after being fully discharged, the event will be recorded.
Time Frame: From the time of consent until 30 days post-operatively
Measure: Count of Participants; unit: Participants
Arm/Group | Acetaminophen Injectable Product | Sodium Chloride 0.9%, Intravenous
Number analyzed (Participants) | 76 | 78
Participants | 9 | 10

9. Secondary Outcome: Patient Satisfaction
Description: Overall patient satisfaction as well as satisfaction relating to pain management and cost analyses will be measured. These will be measured with a numerical rating scale (NRS) with 0- being worst satisfaction and 10 - best satisfaction.
Time Frame: These measurements will be taken at time of discharge up to 30 days, whichever comes first
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Acetaminophen Injectable Product | Sodium Chloride 0.9%, Intravenous
Number analyzed (Participants) | 76 | 78
score on a scale
  Patient satisfaction score, overall | 10 [9 to 10] | 10 [9 to 10]
  Patient Satisfaction score, pain management | 10 [9 to 10] | 10 [8 to 10]

10. Secondary Outcome: Intensive Care Delirium Screening Checklist (ICDSC)
Description: Number of patients who score greater than a 4 on the 0-8 point ICDSC scale to assess delirium scores. 8 separate levels of signs for delirium assessed (1. altered level of consciousness, 2. inattention, 3. disorientation, 4. hallucination, delusion, or psychosis, 5. psychomotor agitation or retardation, 6. inappropriate speech or mood, 7. sleep-wake cycle disturbance, 8. symptom fluctuation), with 0 points awarded when patient does not exhibit above signs of delirium and 1 point awarded per confirmed sign of delirium. Score then totaled, 0 = normal, 1-3 = subsyndromal delirium, 4-8 = delirium.
Time Frame: The delirium scores will first be measured every 12 hours for 72 hours after surgery.
Measure: Count of Participants; unit: Participants
Arm/Group | Acetaminophen Injectable Product | Sodium Chloride 0.9%, Intravenous
Number analyzed (Participants) | 76 | 78
Participants | 0 | 0

11. Secondary Outcome: Post-operative Nausea
Description: Nausea will be evaluated by nausea score from 0 to 10, with 0 equaling no nausea and 10 equaling the worst nausea imaginable.
Time Frame: These will be evaluated from the time of PACU admission until 72 hours postoperatively.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Acetaminophen Injectable Product | Sodium Chloride 0.9%, Intravenous
Number analyzed (Participants) | 76 | 78
score on a scale
  Nausea score POD 1 (am visit) | 1.13 (2.82) | 0.60 (1.76)
  Nausea score POD 1 (pm visit) | 0.49 (1.54) | 0.92 (2.53)
  Nausea score POD 2 (am visit) | 0.71 (1.97) | 0.75 (2.39)
  Nausea score POD 2 (pm visit) | 0.55 (1.70) | 0.69 (2.36)
  Nausea score POD 3 (am visit) | 0.32 (1.37) | 0.66 (2.18)
  Nausea score POD 3 (pm visit) | 0.56 (1.77) | 0.78 (2.42)

12. Secondary Outcome: Post-operative Emesis
Description: Frequency of emesis and rescue antiemetic requirement will be documented
Time Frame: These will be evaluated from the time of PACU admission until 72 hours postoperatively.
Measure: Count of Participants; unit: Participants
Arm/Group | Acetaminophen Injectable Product | Sodium Chloride 0.9%, Intravenous
Number analyzed (Participants) | 76 | 78
Participants
  Emesis incidence 0-72 hours | 12 | 14
  Antiemetic use | 31 | 45

13. Secondary Outcome: SF-12 Health Survey
Description: Survey to assess patient's overall health (via a combination of mental and physical health assessment) at 30 days post-discharge. Two summary scores are reported from the SF-12 - a mental component score (MCS-12) and a physical component score (PCS-12). The scores may be reported as Z-scores (difference compared to the population average, measured in standard deviations). The United States population average PCS-12 and MCS-12 are both 50 points. The United States population standard deviation is 10 points. So each 10 increment of 10 points above or below 50, corresponds to one standard deviation away from the average
Time Frame: These measurements will take place at 30-days post hospital discharge
Measure: Median (Inter-Quartile Range); unit: Z-scores (difference compared to the pop
Arm/Group | Acetaminophen Injectable Product | Sodium Chloride 0.9%, Intravenous
Number analyzed (Participants) | 76 | 78
Z-scores (difference compared to the pop
  SF 12 Physical score | 38.72 [30.73 to 43.28] | 38.07 [32.56 to 45.85]
  SF 12 Mental score | 54.02 [48.33 to 57.42] | 52.08 [42.66 to 57.88]

ADVERSE EVENTS:
Time Frame: 30 Days
Arm/Group | Acetaminophen Injectable Product | Sodium Chloride 0.9%, Intravenous
All-Cause Mortality (participants affected / at risk) | 0/76 | 0/78
Serious Adverse Events (participants affected / at risk) | 3/76 | 3/78
Other Adverse Events (participants affected / at risk) | 8/76 | 8/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Acetaminophen Injectable Product (N=76) | Sodium Chloride 0.9%, Intravenous (N=78)
Acute Kidney Injury (Renal and urinary disorders) | 2 | 1
Respiratory Depression (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pnemonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Acetaminophen Injectable Product (N=76) | Sodium Chloride 0.9%, Intravenous (N=78)
Pruritis (Skin and subcutaneous tissue disorders) | 2 | 0
Anastomotic Leak (Surgical and medical procedures) | 2 | 2
Urinary Retention (Renal and urinary disorders) | 2 | 3
Prolonged Ileus (Gastrointestinal disorders) | 1 | 2
Pancreatic Leak (Surgical and medical procedures) | 0 | 1
Respiratory Depression (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-05): https://cdn.clinicaltrials.gov/large-docs/71/NCT03198871/Prot_SAP_000.pdf